CLINICAL TRIAL: NCT04543565
Title: Pradefovir Treatment for the Patients With Chronic Hepatitis B Virus Infections: a Multi-center, Double-Blind, Randomized, Positive Control, Phase3 Study
Brief Title: Pradefovir Treatment for the Patients With Chronic Hepatitis B Virus Infections: a Phase3 Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BOJI201939F
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): subject in this group will receive Pradefovir mesylate tablet and the placebo of tenofovir disoproxil fumarate tablet, once daily for 96 weeks
  Interventions: Drug: Pradefovir Mesylate;Placebo of Tenofovir disoproxil fumarate tablet
- Control group (Active Comparator): subject in this group will receive tenofovir disoproxil fumarate tablet and the placebo of Pradefovir mesylate tablet, once daily for 96 weeks.
  Interventions: Drug: Tenofovir disoproxil fumarate tablet;Placebo of Pradefovir Mesylate

INTERVENTIONS:
Drug: Pradefovir Mesylate;Placebo of Tenofovir disoproxil fumarate tablet — Once daily
  Arms: Trial group
Drug: Tenofovir disoproxil fumarate tablet;Placebo of Pradefovir Mesylate — Once daily
  Arms: Control group

SUMMARY:
This is a phase three study to evaluate the safety and efficacy of Pradefovir treatment in chronic hepatitis B patients. Subject will be randomized to Pradefovir group and TDF group at a ratio of 2:1. Treatment duration will be 96w in randomization and followed by 48w in open. The interim analysis will be conducted when all subject completed the first 48-week treatment.

DETAILED DESCRIPTION:
this is a randomized, double-blind, positive drug parallel control, multicenter, phase 3 study .Eligible HBeAg-positive or HBeAg-negative chronic hepatitis B patients will be stratified by historical antiviral treatment (untreated or treated) at the time of screening, and then randomly assigned to Pradefovir mesylate tablet group or tenofovir disoproxil fumarate tablet group at a ratio of 2:1. The proportion of subject with compensatory stage of cirrhosis is no more than 20 percentage. Patients will receive a total of 144 weeks of antiviral treatments, and after 96 weeks of double-blind treatment, all subjects will switch to open mesylate Pradefovir tablets for additional 48 weeks. The first 48 weeks are the core period and the followed 96 weeks are the extension period. Statistical analysis was conducted on the efficacy and safety of the whole trial. (After the completion of 48-week visit of the last one subject, the interim analysis will be conducted. The analysts will be unblinded, while the remaining participants will still be blind.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old, male or female.
* Meets the diagnosis and treatment standards of chronic hepatitis B( HBsAg or HBV DNA positive over 6 months, or diagnosed by liver biopsy.
* For HBeAg positive, HBV DNA equal or over 20000 IU/ml; for HBeAg negative ,HBV DNA equal or over 2000 IU/ml.
* ALT level between 1.2 ULN to 10 UNL.
* Treatment naive or experienced when any nucleos(t)ide analogs or interferons stopped over 6 months.
* Use of effective contraceptive measures if procreative potential exists.
* Written informed consent.

Exclusion Criteria:

* Allergic to study drug,metabolite product or excipient.
* Evidence of hepatic decompensation such as Child-Pugh B or C, with previous gastroesophageal variceal haemorrhage, hepatic encephalopathy, ascites
* Suspected or confirmed hepatocellular carcinoma, or AFP>50μg/L.
* Other liver diseases (such as Chronic alcoholic hepatitis, drug-induced hepatitis, autoimmune liver disease).
* Resistant to antiviral drugs (adefovir or tenofovir).
* Concommitant disease of severe heart, blood, respiratory and central nervous system diseases.
* Chronic kidney diseases, or Ccr<60ml/min at screening.
* Abnormal hematological and biochemical parameters at screening: White blood cell count less than 3.0×109/L，or neutrophil count less than 1.5×109/L，or platelet count less than 80×109/L，or total bilirubin more than 2ULN，or the prolong of PT more than 3s.
* Positive-HCV or positive-HIV.
* Severe bone disease (such as osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, rickets) or multiple fractures.
* History of pancreatitis or malignancy within 5 years (excluding cervical epithelial carcinoma, squamous epithelial carcinoma, or basal cell carcinoma of the skin that was clinically cured within 5 years of diagnosis).
* Plan to receive or have already had an organ transplant.
* Subject with disabilities as prescribed by law (blindness, deafness, deafness, deafness, mental disorders, etc.).
* History of alcohol or drug abuse within the last 1 year.
* Pregnant or lactating women.
* Participated in any clinical trial or taken any IMP (investigational medical product) within 3 months prior to the trial.
* Other cases that could not be enrolled in the judgement of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HBV viral suppression | After 48-week therapy
  proportion of patients with hepatitis B virus(HBV) -DNA undetectable(<29IU/ml)

SECONDARY OUTCOMES:
HBV viral suppression | After therapy of 4, 8, 12, 24, 36, 72, 96, 144 weeks
  proportion of patients with hepatitis B virus(HBV) -DNA undetectable(<29IU/ml)
HBV viral suppression | After therapy of 4, 8, 12, 24, 48, 36, 72, 96, 144 weeks
  proportion of patients with hepatitis B virus(HBV) -DNA undetectable(<20IU/ml)
The reduction of HBV DNA load | at week 4, 8, 12, 24, 36, 48, 72, 96, 144
  the change of HBV DNA load from baseline
ALT normalization | After therapy of 4, 8, 12, 24, 48, 36, 72, 96, 144 weeks
  proportion of patients with ALT normalization

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Dr., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China